CLINICAL TRIAL: NCT02105649
Title: CALF MUSCLE STRENGTH AND STANDING EFFICIENCY IN CHILDREN WITH SPASTIC DIPLEGIA: A RANDOMIZED CONTROLLED TRIAL
Brief Title: Calf Muscle Strength and Standing Efficiency in Children With Spastic Diplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Elsayed Elnahhas, assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12345
Record Dates: First submitted 2014-04-03; First posted 2014-04-07 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; standing; strengthening
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- calf muscle strengthenig group (Experimental): experimental group
  will receive the same selected physical therapy program in addition to manual and mechanical strengthening exercises and electrical stimulation program for calf muscles of both lower limbs.
  Interventions: Other: Strengthening exercise + Electrical stimulation of calf muscle; Other: selected physical therapy program
- No calf muscle strengthening group (Other): control group
  will receive only the selected physical therapy program
  Interventions: Other: selected physical therapy program

INTERVENTIONS:
Other: Strengthening exercise + Electrical stimulation of calf muscle
  Arms: calf muscle strengthenig group
Other: selected physical therapy program

SUMMARY:
It will be hypothesized that strengthening the calf muscles will improve standing efficiency in children with spastic diplegia.

ELIGIBILITY:
Inclusion Criteria:

* Children age will be ranging between 2 and 4 years.
* They are classified at level III by GMFCS-ER, i.e. they can stand with minimal support.
* Full mobile lower limbs joints.
* Children with mild and moderate spasticity ( i.e. grade 1 and 2, according to Modified Ashworth Scale).

Exclusion Criteria:

* Children with severe spasticity ( i.e. grade 4, according to Modified Ashworth Scale).
* Fixed deformities.
* Uncontrolled seizures.

Ages: 2 Years to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2014-07 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure | 2 months

SECONDARY OUTCOMES:
Ultrasonography | 2 months
  To measure calf muscle thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Giza Governorate, Egypt

REFERENCES:
- [Background] Wiley ME, Damiano DL. Lower-extremity strength profiles in spastic cerebral palsy. Dev Med Child Neurol. 1998 Feb;40(2):100-7. doi: 10.1111/j.1469-8749.1998.tb15369.x. PMID 9489498